CLINICAL TRIAL: NCT04178057
Title: An Open-label, Dose-escalated, Phase I Clinical Trial to Assess the Safety, Tolerability and Pharmacokinetic Profiles of GB222 in Chinese Patients With Relapsed/Progressive High-grade Glioma
Brief Title: Phase I Clinical Study of GB222 to Evaluate the Safety, Tolerability and PK Profiles.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GENOR GB222-003; V2.1
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GB222 3mg/kg (Experimental): GB222 3mg/kg
  Interventions: Biological: GB222 3mg/kg
- GB222 5mg/kg (Experimental): GB222 5mg/kg
  Interventions: Biological: GB222 5mg/kg
- GB222 7.5mg/kg (Experimental): GB222 7.5mg/kg
  Interventions: Biological: GB222 7.5mg/kg
- GB222 10mg/kg (Experimental): GB222 10mg/kg
  Interventions: Biological: GB222 10mg/kg

INTERVENTIONS:
Biological: GB222 3mg/kg — Injection, strength 100mg/bottle, intravenous infusion, 3mg/kg, dose escalation; After it is tolerated, 2 weeks/per time, combines use of chemotherapeutic agents is allowed after 3 months until disease progression, death, intolerable toxic reactions, withdrawal of informed consent form, loss to follow-up, death or study conclusion; low dose group.
  Other Names: Recombinant humanized antivascular endothelial growth factor monoclonal antibody injection
  Arms: GB222 3mg/kg
Biological: GB222 5mg/kg — Injection, strength 100mg/bottle, intravenous infusion,5mg/kg, dose escalation; After it is tolerated, 2 weeks/per time, combines use of chemotherapeutic agents is allowed after 3 months until disease progression, death, intolerable toxic reactions, withdrawal of informed consent form, loss to follow-up, death or study conclusion; intermediate dose group 1.
  Other Names: Recombinant humanized antivascular endothelial growth factor monoclonal antibody injection
  Arms: GB222 5mg/kg
Biological: GB222 7.5mg/kg — Injection, strength 100mg/bottle, intravenous infusion,7.5mg/kg, dose escalation; After it is tolerated, 2 weeks/per time, combines use of chemotherapeutic agents is allowed after 3 months until disease progression, death, intolerable toxic reactions, withdrawal of informed consent form, loss to follow-up, death or study conclusion; intermediate dose group 2.
  Other Names: Recombinant humanized antivascular endothelial growth factor monoclonal antibody injection
  Arms: GB222 7.5mg/kg
Biological: GB222 10mg/kg — Injection, strength 100mg/bottle, intravenous infusion,10mg/kg, dose escalation; After it is tolerated, 2 weeks/per time, combines use of chemotherapeutic agents is allowed after 3 months until disease progression, death, intolerable toxic reactions, withdrawal of informed consent form, loss to follow-up, death or study conclusion; high dose group.
  Other Names: Recombinant humanized antivascular endothelial growth factor monoclonal antibody injection
  Arms: GB222 10mg/kg

SUMMARY:
This study is designed to assess the safety and tolerability, pharmacokinetic profiles, immunogenicity of GB222 in Chinese patients with relapsed/progressive high-grade glioma; moreover, changes in cerebral edema, changes in KPS score from baseline, objective response rate (ORR), 4-month progression-free survival (PFS), overall survival (OS)will be evaluated. The dose reduction of hormone during continuous administration period will be observed.

ELIGIBILITY:
Inclusion Criteria:

The patients can be enrolled only if they meet the following all inclusion criteria:

1. Age ≥ 18 years, male or female;
2. Understand the study procedures and contents, and voluntarily sign the written informed consent form;
3. Histologically or cytologically confirmed advanced high-grade glioma which failed respond to conventional treatment and is unsuitable to receive multidisciplinary treatment, WHO grades III-IV;
4. Disease progression (recurrence) after first-line treatment including surgery, radiotherapy and temozolomide chemotherapy;
5. MRI confirmed tumor progression (within 14 days before the administration of investigational product);
6. KPS score ≥50;
7. Life expectancy≥3 months;
8. The resection of relapsed brain tumors is performed at least 4 weeks before the use of investigational products, or sereotactic mamography biopsy of brain tumors is performed at least 2 weeks before the use of investigational products;
9. The radiotherapy is performed at least 12 weeks before the use of investigational products, unless that the size increased of relapsed tumor is larger than that of the site received radiotherapy or histologically confirmed tumor progression;
10. The chemotherapy is completed at least 4 weeks before the use of investigational products;
11. At least one measurable and evaluable tumor lesion (in accordance with RANO criteria);
12. Prior to the use of investigational product, all adverse reactions related to the previous treatment must recover to the level specified in the inclusion criteria, grade 0 or 1 (the following is excluded -including but not limited to alopecia, laboratory parameters in the inclusion criteria and common lymphocytopenia after temozolomide treatment);
13. The investigational products can be used after 5 half-lives of other previously used investigational products, after 4 weeks of cytotoxic agents (23 days for temozolomide, 6 weeks for nitrosoureas) and after 4 weeks of monoclonal antibodies (or 5 half-lives, whichever is longer);
14. Subjects who have no serious hematological, cardiopulmonary, hepatorenal disease, hemoglobin (Hb) ≥9g/dl, white blood cell count ≥3.5×109/L, neutrophil ≥1.5×109/L, platelet≥100×109/L; serum creatinine (Cr) ≤1.5xULN or calculated value of creatinine clearance *≥50mL/min; urine protein < 2+ or less than 1.0g/L (if urine protein in routine urine test is ≥2+ or 1.0g/L at baseline, quantitative test of 24h urinary protein shall be performed. If it is < 1g/24 hours, the subjects can be enrolled); total bilirubin < 1.0xULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5xULN; international normalized ratio (INR) ≤1.0xULN, and prothrombin time (PT) and activated partial thromboplastin time (APTT)≤1.0xULN;
15. Females of child-bearing potential have negative pregnancy test; males or females agree to adopt medically confirmed effective contraceptive measures during the entire study period and within 6 months after the end of this study.
16. Patients can receive follow-up visits as scheduled, well communicate with the investigators and complete the study as required by the study. *Ccr for males=(140-age) × body weight (kg)/(72×Scr (mg/dl)); or Ccr for females=[(140-age)×body weight (kg)]/[85×Scr (mg/dl)]

Exclusion criteria:

The subjects are not allowed to participate in this clinical study if they meet any of the following criteria:

1. Subjects with brain neoplasms which occur in brain stem;
2. Subjects with diffuse meningeal dissemination;
3. Subjects who previously had other malignancies (excluding cured cervical carcinoma in situ and skin basal cell carcinoma) are not allowed to participate in the study unless he/she completely relieved at least 2 years before being enrolled in this study and requires no other treatment now or during the study period.
4. Subjects who have active, known or suspected autoimmune diseases;
5. Subjects who received treatment with systemic immunosuppressive therapies within 6 months before the use of investigational products;
6. Subjects who received large dose of systemic glucocorticoids within 2 weeks before the use of investigational products, which is equivalent to dexamethasone >4.1mg/d or equivalent dose, administration for 3 continuous days[3].
7. Subjects who previously received isotopic radiotherapy, implanted chemotherapy, stereotactic radiotherapy or local injection or convection-enhanced delivery (CED);
8. The medical history or test results showing thrombotic diseases within 6 months before enrollment;
9. Subjects who received larger surgical procedures, experienced significant trauma, or expected to receive major surgery during the study treatment period within 4 weeks before the use of investigational products;
10. Subjects who received minor surgical procedures (including cannulation) within 48 hours before the use of the first monoclonal antibody and are considered to have bleeding tendency at the discretion of the investigator;
11. Subjects who currently or recently (within 10 days before the first dose of monoclonal antibody) used aspirin (>325mg/day) or other non-steroidal anti-inflammatory drugs (NSAIDs) which are known to inhibit platelet function;
12. Subjects who currently or recently (within 10 days before the first dose of monoclonal antibody) are treated with whole dose of oral or parenteral anticoagulants or thrombolytic therapies;
13. The medical history or test results showing hereditary bleeding tendency or coagulation disorders, thus increasing the risks of bleeding;
14. Patients with complicated serious internal diseases, including uncontrolled diabetes mellitus, active gastrointestinal ulcer, active bleeding etc.;
15. Uncontrolled hypertension (systolic blood pressure >140 mmHg and/or diastolic pressure > 90 mmHg);
16. Patients who previously have hypertensive crisis or hypertensive encephalopathy;
17. Subjects with clinical significant (e.g., active) cerebrovascular diseases, e.g., cerebrovascular accident (CVA) or transient ischemic attack (TIA) (≤6 months before enrollment), myocardial infarction (≤6 months before enrollment), unstable angina pectoris, congestive heart failure (New York Heart Association grade III or above), subjects who require drug therapies during the study period which may interfere study treatment, or subjects with serious arrhythmia which cannot be controlled by drugs;
18. Subjects with significant vascular diseases within 6 months before the use of investigational products (including but not limited to aortic aneurysm requiring repair surgery or recent artery thrombosis);
19. Subjects with non-cured wound, active peptic ulcer or fracture;
20. Subjects who are diagnosed with tracheoesophageal fistula;
21. Subjects who have medical history of abdominal fistula, gastrointestinal perforation or intraperitoneal abscess;
22. Subjects who have active infection (≥CTCAE grade 2);
23. Previously or currently suffering from active pulmonary tuberculosis (TB) infection;
24. Any of the following is positive: hepatitis C antibody (HCV-Ab), acquired immunodeficiency syndrome antibody (Anti-HIV) and anti-treponema pallidum antibody (TP-Ab);
25. Positive hepatitis B surface antigen (HBsAg) and peripheral blood hepatitis B virus deoxyribonucleic acid (HBV-DNA) >103 copies/L, if HBV-DNA titer test <103 copies/L, and the investigator considers that chronic hepatitis B is stable and cannot increase the risks, the subjects can be enrolled;
26. Patients who had used other investigationsl drugs within 28 days before the use of this investigational drug or within 5 half-lives of the previous investigational drugs (whichever is longer) or had used investigational medical device within 28 days;
27. Patients who received any anti-infection vaccines (e.g. influenza vaccine, varicella vaccine etc.) within 4 weeks before enrollment;
28. Subjects with drug addiction or alcohol addiction (i.e., weekly alcohol consumption > 14 units, one unit of alcohol=360ml of beer or 45ml 40% liquor or 150 mL of wine)
29. Subjects with interstitial lung disease and clinical symptoms;
30. Subjects with peripheral neuropathy ≥ CTCAE grade 2
31. Subjects who are known to be allergic to anti-VEGF monoclonal antibody or any of its excipients, or subjects who are known to have medical history of allergic diseases or allergic constitution;
32. Subjects who received anti-VEGF monoclonal antibody or similar products before the study;
33. Pregnant and lactating women;
34. Patients who have poor compliance, self-care disability and cannot guarantee to follow the protocol requirements;
35. Subjects who are considered unsuitable for participating in this study for various reasons at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity, DLT | up to 28 days
  Dose-limiting toxicity, DLT
Maximum Tolerated Dose, MTD | up to 28 days
  Maximum Tolerated Dose, MTD
Serious Adverse Effect, SAE | up to 28 days
  Serious Adverse Effect, SAE
Adervse Effect, AE | up to 28 days
  Adervse Effect, AE

SECONDARY OUTCOMES:
Cmax | up to 28 days
  Cmax
AUC 0-t | up to 28 days
  AUC 0-t
AUC (0- ∞) | up to 28 days
  AUC (0- ∞)
Tmax | up to 28 days
  Tmax
T 1/2 | up to 28 days
  T 1/2
CL | up to 28 days
  CL
Antidrug Antibody, ADA | through study completion, an average of 2 year
  Antidrug Antibody, ADA
Objective Response Rate, ORR | through study completion, an average of 2 year
  Objective Response Rate, ORR
Progress-free Survial, PFS | through study completion, an average of 2 year
  Progress-free Survial, PFS
Overall Survial, OS | through study completion, an average of 2 year
  Overall Survial, OS

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Li, Ph.D, Principal Investigator — Beijing Tiantan Hospital of Capital Medical University
Locations (1):
- Beijing Tiantan Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No